CLINICAL TRIAL: NCT01906853
Title: A Randomised, Controlled Trial to Determine if BCG Immunisation at Birth Reduces Allergy and Infection in Infants
Brief Title: Melbourne Infant Study - Bacille Calmette Guérin (BCG) for Allergy & Infection Reduction
Acronym: MIS BAIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Mercy Hospital for Women, Australia (Other); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BCG12/01; 1051228 (Other Grant/Funding Number: National Health and Medical Research Council (NHMRC))
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Allergy; Eczema; Respiratory Tract Infections
Keywords: BCG; Bacille Calmette Guérin; Allergy; Immunity; Immune response; Vaccine; Infants; Children; Infection
MeSH Terms: conditions — Hypersensitivity; Eczema; Respiratory Tract Infections; Infections | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No BCG (No Intervention): No BCG
- BCG (Experimental): Mycobacterium bovis BCG (Bacille Calmette Guérin) vaccine, Danish Strain 1331
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: BCG
  Other Names: BCG vaccine - Denmark strain; BCG Denmark; Statens Serum Institute BCG vaccine; Mycobacterium bovis BCG (Bacille Calmette Guérin), Danish Strain 1331
  Arms: BCG

SUMMARY:
1. To determine if BCG immunisation at birth, compared to no BCG immunisation, leads to a reduction in measures of allergy and infection in the first 12 months of life.
2. To evaluate the immunological mechanisms underlying the non-specific effects of BCG by comparing markers of immunity between the BCG and non-BCG groups.

DETAILED DESCRIPTION:
There has been a dramatic rise in allergic diseases worldwide since the 1980s. Asthma rates increased first, followed by eczema, allergic rhinitis and, more recently, food allergy - especially in infants and young children. In Australia, the prevalence of allergic disease is particularly high: up to 30% of children are affected, and eczema and asthma are among the most common chronic diseases of childhood.

Preventing allergic disease by an immunomodulatory intervention early in life would be a major advance with significant implications for individual health and public health resources. Bacillus Calmette-Guérin (BCG) immunisation is a potential intervention with an established safety profile. This vaccine has powerful non-specific effects on the cellular immune response that potentially prime host immunity away from an allergic pathway. Observational data and one small randomised controlled trial (RCT) suggest that BCG immunisation at birth leads to a substantial reduction in allergic disease - however, there is an absence of level 1 evidence.

ELIGIBILITY:
Inclusion criteria:

* Less than 10 days old;
* English speaking mother;
* An informed consent form must be signed and dated by their parent(s) or legally acceptable representative after the nature of the study has been explained and prior to any study assessments/procedures;
* The infant's mother has screened negative for HIV during this pregnancy;
* Born no earlier than eight weeks before estimated date of delivery;
* Birth weight >1500g.
* The legal guardian expects to be able to complete four online/phone questionnaires over the infant's first 12 months of life and for the infant to be available for skin prick testing at RCH between 12-16 months of age.

Exclusion criteria:

* Any indication for BCG immunisation in the first 12 months of life including:

  * likely travel to a high tuberculosis (TB) incidence country in the first year of life.
  * Aboriginal and Torres Strait Islander babies living in parts of Australia where the incidence of TB is higher
  * newborn babies, if either parent has leprosy or a family history of leprosy
  * newborn in contact with a patient with TB.
* Known or suspected HIV infection
* Treatment with corticosteroids or other immunosuppressive therapy, including monoclonal antibodies against tumour necrosis factor-alpha (TNF-alpha) (e.g. infliximab, etanercept, adalimumab).
* Born to a mother treated with bDMARDS (e.g. TNF-alpha blocking monoclonal antibodies) in the 3rd trimester;
* Congenital cellular immunodeficiencies including specific deficiencies of the interferon gamma pathway;
* Malignancies involving bone marrow or lymphoid systems;
* Serious underlying illness including severe malnutrition;
* Medically unstable;
* Generalised septic skin disease and skin conditions such as eczema, dermatitis and psoriasis;
* Significant febrile illness;
* Mother immunosuppressed;
* Family history of immunodeficiency;
* Consanguineous parents;
* Multiple births more than twins.

Max Age: 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1272 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2025-02 (Actual)

PRIMARY OUTCOMES:
Atopic sensitisation measured by skin prick test (SPT) | 1 year of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to one or more of a panel of food and aeroallergens
Atopic sensitisation measured by skin prick test (SPT) | 5 years of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to one or more of a panel of food and aeroallergens
Lower respiratory tract infection (LRTI) | 0-12 months
  Measured by parent report
Lower respiratory tract infection (LRTI) hospital admissions | 0-5 years of age
  Proportion of participants with ≥1 hospital admission for LRTI reported by parent
Eczema ever | 0-12 months
  Proportion of participants with eczema measured by Williams' UK diagnostic criteria using parental report of symptoms
Eczema ever | 0-5 years of age
  Proportion of participants with eczema measured by Williams' UK diagnostic criteria using parental report of symptoms
Current asthma | 5 years of age
  Using ISAAC definitions
Asthma ever | 5 years of age
  Using ISAAC definitions

SECONDARY OUTCOMES:
Clinical food allergy | 1 year of age
  Proportion of participants with challenge-proven food allergy OR convincing history of food allergy in participants with a SPT wheal diameter ≥2 mm greater than negative control at 15 min to one or more of a panel of food allergens
Clinical food allergy | 5 years of age
  Proportion of participants with challenge-proven food allergy OR convincing history of food allergy in participants with a SPT wheal diameter ≥2 mm greater than negative control at 15 min to one or more of a panel of food allergens
Atopic sensitisation measured by SPT using a more stringent cut-off | 1 year of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥3 mm greater than negative control at 15 min to one or more of a panel of food allergens and aeroallergens
Atopic sensitisation measured by SPT using a more stringent cut-off | 5 years of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥3 mm greater than negative control at 15 min to one or more of a panel of food allergens and aeroallergens
Atopic sensitisation to multiple allergens measured by SPT | 1 year of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to two or more of a panel of food allergens and aeroallergens
Atopic sensitisation to multiple allergens measured by SPT | 5 years of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to two or more of a panel of food allergens and aeroallergens
Parent report of food allergy | 0-12 months of age
  Proportion of participants with an allergic reaction to any food reported by parent
Parent report of food allergy | 0-5 years of age
  Proportion of participants with an allergic reaction to any food reported by parent
Egg sensitisation | 1 year of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to egg allergen
Egg sensitisation | 5 years of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to egg allergen
Egg allergy | 1 year of age
  Proportion of participants with a challenge-proven egg allergy OR convincing history of egg allergy in participants with a SPT wheal diameter ≥2 mm greater than negative control at 15 min to egg
Egg allergy | 5 years of age
  Proportion of participants with a challenge-proven egg allergy OR convincing history of egg allergy in participants with a SPT wheal diameter ≥2 mm greater than negative control at 15 min to egg
Atopic wheeze | 1 year of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to one or more of a panel of food and aeroallergens together with parent-reported wheeze
Atopic wheeze | 5 years of age
  Proportion of participants with a positive SPT defined as wheal diameter ≥2 mm greater than negative control at 15 min to one or more of a panel of food and aeroallergens together with parent-reported wheeze
Lower respiratory tract infection (LRTI) | Prior to first Diphtheria, Tetanus, Pertussis (DTP) vaccination
  Proportion of participants with ≥1 episode of LRTI, by parental report
Lower respiratory tract infection (LRTI) | 0-5 years of age
  Proportion of participants with ≥1 episode of LRTI, by parental report
Rate of lower respiratory tract infection (LRTI) | 0-12 months
  Number of clinical episodes of LRTI, by parental report
Rate of lower respiratory tract infection (LRTI) | Prior to first DTP vaccination
  Number of clinical episodes of LRTI, by parental report
Rate of lower respiratory tract infection (LRTI) | 0-5 years of age
  Number of clinical episodes of LRTI, by parental report
Infections | 0-12 months
  Hospital admissions for any infection by parental report
Infections | Prior to first DTP vaccination
  Hospital admissions for any infection by parental report
Infections | 0-5 years of age
  Hospital admissions for any infection by parental report
Hospitalisation for respiratory tract infection (RTI) | 0-12 months of age
  Proportion of participants with ≥1 hospital admission for a RTI, by parent report
Hospitalisation for respiratory tract infection (RTI) | Prior to first DTP vaccination
  Proportion of participants with ≥1 hospital admission for a RTI, by parent report
Hospitalisation for respiratory tract infection (RTI) | 0-5 years of age
  Proportion of participants with ≥1 hospital admission for a RTI, by parent report
Rate of any infection | 0-12 months of age
  Number of clinical episodes of where an infant had symptoms of: wheeze, rattle/rattly chest, fever, runny/blocked nose, cough, or diarrhoea (with vomiting), by parent report
Rate of any infection | Prior to first DTP vaccination
  Number of clinical episodes of where an infant had symptoms of: wheeze, rattle/rattly chest, fever, runny/blocked nose, cough, or diarrhoea (with vomiting), by parent report
Rate of upper respiratory tract infection (URTI) | 0-12 months of age
  Number of clinical episodes of upper respiratory tract infections, by parent report
Rate of upper respiratory tract infection (URTI) | Prior to first DTP vaccination
  Number of clinical episodes of upper respiratory tract infections, by parent report
Rate of fever | 0-12 months of age
  Number of clinical episodes of fever, by parent report
Rate of fever | Prior to first DTP vaccination
  Number of clinical episodes of fever, by parent report
Diarrhoea | 0-12 months of age
  Proportion of participants with ≥1 episodes of diarrhoea
Diarrhoea | Prior to first DTP vaccination
  Proportion of participants with ≥1 episodes of diarrhoea
Rash with fever | 0-12 months of age
  Proportion of participants with ≥1 episodes of rash with fever
Rash with fever | Prior to first DTP vaccination
  Proportion of participants with ≥1 episodes of rash with fever
Eczema ever | 0-12 months of age
  Proportion of participants with eczema measured by a combined eczema measure
Eczema ever | 0-5 years of age
  Proportion of participants with eczema measured by a combined eczema measure
Eczema | 0-12 months
  Proportion of clinician-diagnosed eczema, by parental report
Eczema | 0-5 years of age
  Proportion of clinician-diagnosed eczema, by parental report
Eczema onset | 0-12 months
  Age of onset of eczema, by parental report
Eczema onset | 0-5 years of age
  Age of onset of eczema, by parental report
Eczema severity | 0-12 months
  Measured by parental report (POEM score)
Eczema severity | 0-12 months
  Measured by clinical assessment (SCORAD)
Eczema severity | 0-12 months
  Eczema medication use, by parental report
Eczema severity | 0-5 years of age
  Measured by parental report (POEM score)
Eczema severity | 0-5 years of age
  Measured by clinical assessment (SCORAD)
Eczema severity | 0-5 years of age
  Eczema medication use, by parental report
Asthma severity | 4 years of age
  Measured by asthma control test (ACT), by parental/participant report
Asthma severity | 5 years of age
  Measured by asthma control test (ACT), by parental/participant report
Asthma severity | 2-5 years of age
  Hospital admissions for asthma, by parental report
Laboratory measures of the immune response | Time Frame: 0-5 years of age

OTHER OUTCOMES:
Effect of sex on the non-specific effects BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of maternal BCG on the non-specific effects BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of presence or absence BCG scar on the non-specific effects of BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of timing of BCG administration on the non-specific effects BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of mode of delivery on the non-specific effects BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of family history of allergy on the allergy and eczema outcomes | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of season of birth on the non-specific effects BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Effect of hepatitis B vaccine timing birth on the non-specific effects BCG | 0-12 months and 0-5 years of age
  Sub-group analysis
Meta-analysis | 36 months
  Joint meta-analysis with data from the Danish Calmette study (NCT01694108)
Morbidity | 0-12 months of age
  Hospital admissions for any reason by parental report
Morbidity | 0-5 years of age
  Hospital admissions for any reason by parental report

CONTACTS AND LOCATIONS:
Overall Officials: Prof Nigel Curtis, MBBS DCH DTM&H MRCP FRCPCH PhD, Principal Investigator — Murdoch Children's Research Institute, Royal Children's Hospital, University of Melbourne
Locations (2):
- Australia (2):
  - Mercy Hospital for Women, Heidelberg, Victoria
  - Royal Children's Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Khazaei Y, Kodikara S, Butler CA, Messina NL, Le Cao KA, Dashper SG, Silva MJ. Development and validation of diagnostic and prognostic prediction tools for dental caries in young children through prospective and cross-sectional observational studies: a protocol. BMJ Open. 2025 Oct 5;15(10):e105145. doi: 10.1136/bmjopen-2025-105145. PMID 41047269
- [Derived] Pittet LF, Forbes EK, Donath S, Francis KL, Gardiner K, Flanagan KL, Ponsonby AL, Robins-Browne R, Shann F, South M, Vuillermin P, Casalaz D, Curtis N, Messina NL; Melbourne Infant Study: BCG for Allergy and Infection Reduction (MIS BAIR) Group. Neonatal BCG vaccination to prevent asthma: Results from the MIS BAIR randomized controlled trial. Pediatr Allergy Immunol. 2025 Jun;36(6):e70110. doi: 10.1111/pai.70110. PMID 40464744
- [Derived] Messina NL, Gardiner K, Pittet LF, Forbes EK, Francis KL, Freyne B, Zufferey C, Abruzzo V, Morison C, Turner H, Allen KJ, Flanagan KL, Ponsonby AL, Robins-Browne R, Shann F, Vuillermin P, Donath S, Casalaz D, Curtis N; Melbourne Infant Study: BCG for Allergy and Infection Reduction (MIS BAIR) Group. Neonatal BCG Vaccination for Prevention of Allergy in Infants: The MIS BAIR Randomised Controlled Trial. Clin Exp Allergy. 2024 Sep;54(9):682-693. doi: 10.1111/cea.14537. Epub 2024 Jul 14. PMID 39004434
- [Derived] Pittet LF, Messina NL, Gardiner K, Freyne B, Abruzzo V, Morrison C, Vuillermin P, Allen KJ, Ponsonby AL, Robins-Browne R, Shann F, Flanagan KL, Donath S, Casalaz D, Phillips R, Curtis N. Discordance Between Diagnosis Tools for Assessing Eczema in Infants: A Challenge for Intervention Trials. Dermatitis. 2022 May-Jun 01;33(3):207-214. doi: 10.1097/DER.0000000000000842. Epub 2022 Feb 16. PMID 35170523
- [Derived] Pittet LF, Messina NL, Gardiner K, Freyne B, Abruzzo V, Francis KL, Morrison C, Zufferey C, Vuillermin P, Allen KJ, Ponsonby AL, Robins-Browne R, Shann F, Flanagan KL, Phillips R, Donath S, Casalaz D, Curtis N. Prevention of infant eczema by neonatal Bacillus Calmette-Guerin vaccination: The MIS BAIR randomized controlled trial. Allergy. 2022 Mar;77(3):956-965. doi: 10.1111/all.15022. Epub 2021 Aug 9. PMID 34309859
- [Derived] Cirovic B, de Bree LCJ, Groh L, Blok BA, Chan J, van der Velden WJFM, Bremmers MEJ, van Crevel R, Handler K, Picelli S, Schulte-Schrepping J, Klee K, Oosting M, Koeken VACM, van Ingen J, Li Y, Benn CS, Schultze JL, Joosten LAB, Curtis N, Netea MG, Schlitzer A. BCG Vaccination in Humans Elicits Trained Immunity via the Hematopoietic Progenitor Compartment. Cell Host Microbe. 2020 Aug 12;28(2):322-334.e5. doi: 10.1016/j.chom.2020.05.014. Epub 2020 Jun 15. PMID 32544459
- [Derived] Messina NL, Gardiner K, Donath S, Flanagan K, Ponsonby AL, Shann F, Robins-Browne R, Freyne B, Abruzzo V, Morison C, Cox L, Germano S, Zufferey C, Zimmermann P, Allen KJ, Vuillermin P, South M, Casalaz D, Curtis N. Study protocol for the Melbourne Infant Study: BCG for Allergy and Infection Reduction (MIS BAIR), a randomised controlled trial to determine the non-specific effects of neonatal BCG vaccination in a low-mortality setting. BMJ Open. 2019 Dec 15;9(12):e032844. doi: 10.1136/bmjopen-2019-032844. PMID 31843845
- [Derived] Zimmermann P, Perrett KP, van der Klis FR, Curtis N. The immunomodulatory effects of measles-mumps-rubella vaccination on persistence of heterologous vaccine responses. Immunol Cell Biol. 2019 Jul;97(6):577-585. doi: 10.1111/imcb.12246. Epub 2019 Mar 28. PMID 30791143